CLINICAL TRIAL: NCT01575262
Title: The Physical Activity Loyalty Card Scheme: A Randomised Controlled Trial to Encourage Physical Activity
Brief Title: The Physical Activity Loyalty Card Scheme
Acronym: PAL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Prof Frank Kee, Professor, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: PAL-v1
Record Dates: First submitted 2012-04-10; First posted 2012-04-11 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Health Behavior; Physical Activity
Keywords: behaviour change; incentives; nudging; physical activity; self-monitoring
MeSH Terms: conditions — Health Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Incentive (Experimental): Participants use their PAL card to self-monitor physical activity levels (intrinsic motivation) and minutes of physical activity were converted to points (1 minute of physical activity = 1 point; capped at 30 points per day) over the 12-week intervention period. Points are redeemed for rewards (extrinsic motivation) at week 6 and week 12.
  Interventions: Behavioral: Non-cash incentives
- No Incentive (Active Comparator): Participants used their PAL card to self-monitor their physical activity levels (intrinsic motivation) over the 12-week intervention period but do not collect points or earn rewards.
  Interventions: Behavioral: Self-monitoring physical activity levels

INTERVENTIONS:
Behavioral: Non-cash incentives — Participants used their PAL card to self-monitor physical activity levels (intrinsic motivation) and minutes of physical activity were converted to points (1 minute of PA = 1 point; capped at 30 points per day) over the 12-week intervention period. Points were redeemed for rewards (extrinsic motivation) at week 6 and week 12.
  Arms: Incentive
Behavioral: Self-monitoring physical activity levels — For those in the 'No Incentive' arm, participants used their PAL card to self-monitor their physical activity levels but did not collect points or earn rewards.
  Arms: No Incentive

SUMMARY:
The purpose of this study is to investigate the effectiveness of using incentives to encourage adults to be physically active.

DETAILED DESCRIPTION:
The investigators developed the Physical Activity Loyalty Card (PAL) Scheme which integrates a novel physical activity tracking system with web-based monitoring and nudge initiatives. The tracking system used Near-Field Communication (NFC) technology and a "loyalty card" (PAL Card) which contained a passive Radio Frequency Identification (RFID) tag. Sensors were placed along footpaths in the outdoor environment, in the gym and exercise studio, and participants scanned their PAL card at the sensor when doing physical activity (e.g. walking). A transaction (card ID, sensor ID, and timestamp) was recorded and sent via SMS to a secure data centre. Participants logged onto a personal account on the study website (www.palcard.co.uk) and received real-time feedback on various aspects of their physical activity including minutes, distance and calories expended.

ELIGIBILITY:
Inclusion Criteria:

* males and females
* aged 18-65 years old
* able to complete 15 minutes of moderate intensity physical activity
* based at least 4 days per week (and 6 hours per day) at worksite

Exclusion Criteria:

* advised by General Practitioner not to participate in exercise

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2011-03; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Physical activity | baseline, week 12 and 6 months
  change in moderate-vigorous physical activity (MVPA)measured using the Global Physical Activity Questionnaire (GPAQ); MVPA using an objective physical activity measure (physical activity tracking system)

SECONDARY OUTCOMES:
SF-8 | baseline, week 12 and 6 months
  health
Euroqol 5D | baseline, week 12 and 6 months
  Quality of life
Physical Activity Self-Efficacy Scale | baseline, week 12 and 6 months
  Physical activity self-efficacy
Work absenteeism | baseline, week 12 and 6 months
  Number of sick days from work
Exit questionnaire | week 12
  Participant satisfaction with study involvement

CONTACTS AND LOCATIONS:
Overall Officials: Frank Kee, Principal Investigator — Queen's University, Belfast
Locations (1):
- Queen's University Belfast, Belfast, Antrim, United Kingdom